## RELIGIOUSLY INTEGRATED COGNITIVE BEHAVIORAL GROUP THERAPY STUDY PROTOCOL 22.02.2024

| Intervention session | Process | Target Outcome |
|---|---|---|
| Session 1:<br>Introduction | The session started with the group leader and participants introducing themselves to each other. The intervention's theoretical basis (CBT and R-CBT) was outlined. Participants were informed about generalized anxiety disorder (GAD) symptoms, coping strategies, spiritual resources and the materials to be used throughout the program. Group norms were established, and expectations were explored to promote active engagement. Additionally, the use of prayer as a coping mechanism and the spiritual motivational role of intention-setting were discussed as integral components of the intervention framework. | -To develop a strong therapeutic alliance and foster group cohesion -To inform group members about the purpose and structure of therapy -To promote self-reflection through spiritual practices -To facilitate insight into the interaction between faith and psychological processes |
| Session 2<br>Psychoeducation<br>and worry<br>awareness<br>training | In the second session, anxiety and other distressing emotions were explored through a spiritual lens, emphasizing their functional and adaptive aspects. Through religious references, these emotions were normalized as natural components of the human experience. The potential spiritual consequences of emotional excess were discussed, and a conceptual link was drawn between self-awareness in CBT and the religious concept of self-knowledge within a faith-based framework. | -To explore anxiety and distressing emotions from a spiritual perspective - To promote emotional normalization and faith-based self-awareness |
| Session 3<br>Re-evaluation of<br>the usefulness of<br>worry | The session focused on identifying and restructuring core beliefs that contribute to the maintenance of anxiety. These included beliefs such as: "worrying helps solve problems," "worry serves as a motivator," "it protects against negative emotions," "it prevents undesirable outcomes," and "it is a sign of being a responsible or moral person." Particular emphasis was placed on restructuring the belief that worry is helpful for problem-solving, using the Islamic concepts of <i>khawf</i> (fear/awareness of consequences) and <i>raja</i> '(hope/trust in divine mercy) as alternative cognitive anchors. | - To adopt a values-<br>based approach to<br>managing anxiety;<br>-To relinquish the use of<br>anxiety as a tool for<br>control<br>- To prioritize effort over<br>outcome<br>-To develop a balanced<br>sense of responsibility |
| Session 4-5<br>Uncertainty<br>recognition and<br>behavioral<br>exposure | Cognitive patterns that foster negative interpretations of uncertainty were explored, with a focus on recognizing the psychological burden of excessive need for control and certainty. The comforting role of faith in coping with the unknown was highlighted. Irrational thoughts were reframed through a religious-spiritual perspective, and an optimistic outlook toward managing potentially negative outcomes was encouraged. Relevant verses from the Qur'an and Hadiths were referenced to support therapeutic discussions. | To use faith and spirituality as resources for navigating uncertainty |
| Session 6-7<br>Problem-solving<br>training | A shift in perspective from perceiving problems as threats to viewing them as opportunities for growth was facilitated. The therapeutic role of reliance on God ( <i>tawakkul</i> ) in problem-solving was examined. A group discussion was held to explore the concept of <i>tawakkul</i> , clarifying common misconceptions, with scriptural references to Qur'anic verses guiding the discourse. | -To support the<br>development of effective<br>problem-solving<br>strategies aligned with<br>participants' faith,<br>values, and personal<br>goals |
| Session 8<br>Written<br>exposure | In this session, the concept of <i>sabr</i> (patience) was addressed as a rational and functional coping mechanism, rather than a passive or fatalistic stance. Participants' cognitive distortions related to the concept were explored, particularly beliefs that equate patience with passive endurance or suppression of emotions. The role of <i>sabr</i> was emphasized during | -To facilitate a comprehensive understanding of the concept of <i>sabr</i> (patience) |

## RELIGIOUSLY INTEGRATED COGNITIVE BEHAVIORAL GROUP THERAPY STUDY PROTOCOL 22.02.2024

emotionally challenging exercises, especially in managing distress that emerged during written exposure tasks. A clear distinction was made between *sabr* and *tahammul* (mere tolerance), underscoring that *sabr* involves active perseverance with purpose and meaning, while *tahammul* often reflects passive endurance without engagement or growth. The session concluded with practical exercises aimed at illustrating how *sabr* can interrupt the anxiety cycle and be consciously integrated into daily life. Participants were encouraged to view *sabr* not only as a spiritual virtue but also as a cognitively grounded skill that supports emotional regulation, resilience, and long-term psychological well-being.

-To enhance the ability to use *sabr* as a functional coping strategy during exposure and anxiety regulation exercises

## Session 9 Written exposure

To balance the negatively oriented nature of anxiety, a gratitude practice was integrated into the session. Participants explored the meaning of gratitude and discussed how to incorporate it into daily life through interactive activities. The practice was emphasized as a functional tool for enhancing positive cognitive focus and promoting psychological wellbeing.

- To redirect mental focus from negative thoughts to positive experiences - To recognize and
- balance negative cognitive biases
  -To internalize beha
- -To internalize behaviors that support psychological well-being

## Session 10 Relapse prevention

In the final session, homework assignments were reviewed, and participants provided feedback on previous sessions, perceived changes, and the most challenging practices. The entire therapeutic process was evaluated. The group leader addressed potential post-treatment difficulties and discussed, within a scriptural context, the role of effort and the spiritual meaning of making mistakes as a relapse prevention strategy.

- -To foster hope and support relapse prevention
- -To evaluate the therapeutic process and promote closure